CLINICAL TRIAL: NCT02136745
Title: Genomic and Clinical Effects Associated With a Relaxation Response Mind-Body Intervention in Patients With Irritable Bowel Syndrome and Inflammatory Bowel Disease
Brief Title: Effects of Relaxation Response Mind-body Intervention in Patients With IBS and IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Branden Kuo, Dr., Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-000757/19; R01DP000339 (NIH)
Record Dates: First submitted 2014-05-08; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Irritable Bowel Syndrome; Inflammatory Bowel Disease
Keywords: Irritable Bowel Syndrome; Inflammatory Bowel Disease; mind body; intervention; group; Relaxation Response; genomic effects
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Relaxation Response Mind-Body Intervention (Experimental): The Relaxation Response Mind-Body Intervention (RR-MBI) involved a 9-week group program conducted by a nurse practitioner or psychologist skilled in MBI, which included a GI-specific session conducted by a physician. The groups met once weekly for 1.5 hours. The program was multidimensional and included daily elicitation of the RR using a variety of methods (including breath focus, single-pointed focus, imagery, contemplation, yoga, and mindful awareness); cognitive reappraisal skills, health enhancing behaviors, and the promotion of optimism and acceptance. Throughout the course of treatment, participants were asked to elicit the RR at home each day for 15-20 minutes.
  Interventions: Behavioral: Relaxation Response Mind-Body Intervention

INTERVENTIONS:
Behavioral: Relaxation Response Mind-Body Intervention — The Relaxation Response Mind-Body Intervention (RR-MBI) involved a 9-week group program conducted by a nurse practitioner or psychologist skilled in MBI, which included a GI-specific session conducted by a physician. The groups met once weekly for 1.5 hours. Three consecutive, mixed-disorder groups, ranging in size from 10 to 18 participants each. The program was multidimensional and included daily elicitation of the RR using a variety of methods (including breath focus, single-pointed focus, imagery, contemplation, yoga, and mindful awareness); cognitive reappraisal skills, health enhancing behaviors, and the promotion of optimism and acceptance. Throughout the course of treatment, participants were asked to elicit the RR at home each day for 15-20 minutes.

SUMMARY:
In this pilot study, the investigators examined whether a relaxation response mind-body intervention could be effectively delivered to mixed groups of IBS and IBD patients and determined the effects of the intervention on quality of life, inflammatory markers, and gene expression using transcriptional profiling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented IBS (confirmed by the Rome III diagnostic criteria for 6 months) or IBD (upper limit for Harvey-Bradshaw index [HBI] = 20, upper limit of simple clinical colitis activity index [SCCAI] = 18) by their primary care provider or gastroenterologist
* 18-75 years old
* Fluent in English

Exclusion Criteria:

* Patients with IBS were excluded if they had abdominal surgery in the past 5 years (with the exception of appendectomy, cholecystectomy) or documentation of GI motility disorder.
* Patients with IBD were excluded if they used NSAIDS chronically, were on a prednisone dose ≥20 mg/day, or if surgery was anticipated in the 10-weeks following enrollment.
* Current evidence of duodenal ulcer, gastric ulcer, diverticulitis, esophagitis or infectious gastroenteritis, or any acute gastrointestinal process, as well as if concurrent total parental nutrition or tube feeding were being used.
* Recent (within the last 4-weeks) changes in IBS/IBD medications, planned changes in diet, or current use of steroids
* Currently pregnant or attempting to become pregnant
* Currently (>3-weeks) practicing Tai Chi, meditation, yoga, individual mind/body based psychotherapy or counseling,
* Initiated psychotherapy within the last 8-weeks
* Using psychotropic medications (except at stable doses for at least 12-weeks),
* Has an untreated psychiatric disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
IBS Quality of Life | Change from Baseline (week 0), Mid-intervention (week 5), Post-intervention (week 10), and Short-term Follow-up (week 13)
  The IBS Quality of Life (IBS-QOL) is a validated disease-specific instruments to assess the disease-specific impact of the intervention. The IBS-QOL is a self-reported quality of life (QOL) measure containing 34 questions specific to IBS that is used to assess the impact of IBS and its treatment on QOL.
IBS Symptom Severity Index | Change between Baseline (week 0), Mid-intervention (week 5), Post-intervention (week 10), and Short-term Follow-up (week 13)
  The IBS Symptom Severity Index (SSI) is a validated disease-specific instruments to assess the disease-specific impact of the intervention. The IBS SSI is a widely used questionnaire measuring IBS-related pain frequency, severity of pain, bloating, bowel habit dissatisfaction and interference with daily life and extra-colonic symptoms on a visual analogue scale.
IBD Questionnaire | Change between Baseline (week 0), Mid-intervention (week 5), Post-intervention (week 10), and Short-term Follow-up (week 13)
  The IBD Questionnaire (IBD-Q) is a validated disease-specific instruments to assess the disease-specific impact of the intervention. The IBD-Q is designed to measure the effects of inflammatory bowel disease on daily function and quality of life.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Change between Baseline (week 0), Mid-intervention (week 5), Post-intervention (week 10), and Short-term Follow-up (week 13)
  To measure symptoms common to IBS and IBD, the State-Trait Anxiety Inventory (STAI-Y) was administered at each assessment. The STAI is a widely used instrument for measuring anxiety in adults. It differentiates between the temporary condition of "state anxiety" and the more general and long-standing quality of "trait anxiety".
Pain Catastrophizing Scale | Change between Baseline (week 0), Mid-intervention (week 5), Post-intervention (week 10), and Short-term Follow-up (week 13)
  To measure symptoms common to IBS and IBD, the Pain Catastrophizing Scale (PCS) was administered at each assessment. The PCS is widely used to assess cognitive and affective responses to pain and to evaluate pain management program outcomes.
Brief Pain Inventory | Change between Baseline (week 0), Mid-intervention (week 5), Post-intervention (week 10), and Short-term Follow-up (week 13)
  To measure symptoms common to IBS and IBD the Brief Pain Inventory (BPI) was administered at each assessment. The BPI allows patients to rate the severity of their pain (BPI-S) and the degree to which their pain interferes with common dimensions of feeling and function (BPI-I).
erythrocyte sedimentation rate | Change between Baseline (week 0) and Post-intervention (week 10)
  Blood was collected for erythrocyte sedimentation rate (ESR) as measures of inflammation.
C-reactive protein | Change between Baseline (week 0) and Post-intervention (week-10)
  Blood was collected for C-reactive protein (CRP) assays as measures of inflammation.

OTHER OUTCOMES:
Genetic Expression | Change between Baseline (week 0) and Post-Intervention (week 10)
  Blood was collected in PAXgene (Qiagen) tubes for transcriptional expression profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kuo, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kuo B, Bhasin M, Jacquart J, Scult MA, Slipp L, Riklin EI, Lepoutre V, Comosa N, Norton BA, Dassatti A, Rosenblum J, Thurler AH, Surjanhata BC, Hasheminejad NN, Kagan L, Slawsby E, Rao SR, Macklin EA, Fricchione GL, Benson H, Libermann TA, Korzenik J, Denninger JW. Genomic and clinical effects associated with a relaxation response mind-body intervention in patients with irritable bowel syndrome and inflammatory bowel disease. PLoS One. 2015 Apr 30;10(4):e0123861. doi: 10.1371/journal.pone.0123861. eCollection 2015. PMID 25927528